CLINICAL TRIAL: NCT01720732
Title: Lifeline-NET (Narrative Exposure Therapy): A Short-term Treatment for Traumatized Refugees and Asylum Seekers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Konstanz (Other)
Responsible Party: Principal Investigator, Martina Ruf, PhD, University of Konstanz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LL-NET2012
Record Dates: First submitted 2012-08-07; First posted 2012-11-02 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Trauma Treatment; Lifeline NET; Modification of Narrative Exposure Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifeline NET (Experimental): Lifeline-NET (Short Version of NET)
  Interventions: Behavioral: Lifeline NET
- TAU (No Intervention): Treatment as Usual

INTERVENTIONS:
Behavioral: Lifeline NET — Short Version of Narrative Exposure Therapy
  Other Names: LL-NET
  Arms: Lifeline NET

SUMMARY:
Evaluation of a short version of Narrative Exposure Therapy

ELIGIBILITY:
Inclusion Criteria:

* PTSD

Exclusion Criteria:

* Psychotic Disorder,
* Severe Substance Dependence

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2012-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
PTSD | 9 months follow up
  Posttraumatic Stress Disorder Clinician Administered PTSD Scale

SECONDARY OUTCOMES:
Other Symptoms following and related to Trauma, e.g. Depression, Dissociation | 9 months follow up
  Other Symptoms following and related to Trauma, e.g. Depression, Dissociation

OTHER OUTCOMES:
Social functioning, Life Satisfaction, Aggression | 9 months follow up

CONTACTS AND LOCATIONS:
Locations (1):
- University of Konstanz, Konstanz, Germany

REFERENCES:
- [Background] Schauer M, Neuner F, Elbert T (2005/2011): Narrative Exposure Therapy. A Short-Term Intervention for Traumatic Stress Disorders. 2nd Ed. Cambridge/ Göttingen: Hogrefe & Huber Publishers.
- See also: NGO — http://www.vivo.org/